CLINICAL TRIAL: NCT00985374
Title: Multiple Ascending Dose (MAD) Phase Ib/II Study of the mTOR Inhibitor (RAD001) in Combination With the IGF-1R Antagonist (R1507) for the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Multiple Ascending Dose Study of the mTOR Inhibitor (RAD001) in Combination With R1507 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO21884; 2008-005806-38
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Everolimus; RG-1507 monoclonal antibody

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RAD001; Drug: RG1507

INTERVENTIONS:
Drug: RAD001 — 5mg or 10mg po daily
Drug: RG1507 — 16mg/kg iv every 3 weeks

SUMMARY:
This 2 part study will assess the safety, tolerability and efficacy of a combination of oral daily RAD001 and intravenous 3-weekly R1507 in patients with advanced solid tumors. In Part 1 of the study, patients will be enrolled sequentially to receive 5mg by mouth (po) RAD001 daily + 16mg/kg intravenous (iv) R1507 every 3 weeks (level 1) and if tolerated, 10mg po RAD001 daily + 16mg/kg iv R1507 every 3 weeks (level 2).In Part 2 of the study, patients with 1) advanced renal cell cancer and 2) advanced pancreatic neuroendocrine tumors will receive the maximum tolerated dose regimen from Part 1 (5mg or 10mg po RAD001 + 16mg/kg iv R1507). The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* histologically confirmed recurrent or refractory advanced solid tumor (Part 1);
* advanced metastatic renal cell cancer OR advanced metastatic pancreatic neuroendocrine tumors, with evidence of progressive disease (Part 2);
* measurable disease (Part 2);
* ECOG performance status 0-2.

Exclusion Criteria:

* prior treatment with agents acting via inhibition of IGF-IR pathway;
* prior treatment with agents acting via inhibition of mTOR (Part 2);
* untreated CNS metastases;
* current anti-cancer therapy, or radiotherapy or chemotherapy <=4 weeks prior to enrollment;
* other known malignancy requiring treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of RAD001, in combination with R1507 (Part 1 | First 3 week cycle of treatment
Progression-free survival (Part 2) | 24 weeks

SECONDARY OUTCOMES:
Overall objective response rate; duration of response; overall survival | Event driven; monitored throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (2):
  - New York, New York
  - San Antonio, Texas
- Milan, Lombardy, Italy